CLINICAL TRIAL: NCT06337760
Title: YOUNg Adults With Gastro-inteSTinal (GI) and nEuroendocrine canceRs (YOUNGSTER).
Brief Title: YOUNg Adults With Gastro-inteSTinal (GI) and nEuroendocrine canceRs.
Acronym: YOUNGSTER
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1669
Record Dates: First submitted 2024-03-18; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Neuroendocrine Neoplasm; Adenocarcinoma
Keywords: young adult; Gastro-intestinal cancer; Neuroendocrine cancer; molecular analysis; prognostic biomarker
MeSH Terms: conditions — Neuroendocrine Tumors; Adenocarcinoma; Carcinoma, Neuroendocrine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — tumor sample blood sample (optional)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- neuroendocrine neoplasm young patient: Patients aged at diagnosis from18 to 39 years of age with neuroendocrine neoplasm NEN from Gastroenteropancreatic (GEP) or lung/thymus origin
- adenocarcinoma young patient: Patients aged at diagnosis from18 to 39 years of age with carcinoma (without limitations for histologic subtypes) from any primary sites: esophagus, stomach, pancreas, biliary tract, liver, small bowel, colon, rectum, anus and cancer of unknown origin.

SUMMARY:
The objective of the study is to create a common and unique platform for the acquisition of biological samples and, subsequently, the possible identification of predictive and prognostic biomarkers for young adults with gastrointestinal and neuroendocrine cancers.The definition "adolescent and young adults (AYA)" covers a broad group of patients ranging from the upper limit of the paediatric competence to the youngest patients usually considered and treated as adults. However, a well-defined and universally accepted age range is still not established. Young adults with cancer have distinct epidemiological, biological, and clinical characteristics, as well as special medical and psychosocial needs that are often unmet. In consideration of their poor representation in clinical studies, as well as the rarer, albeit increasing, frequency at an epidemiological level, knowledge of the risk factors associated with cancers in young adults is very poor. It is therefore of fundamental importance to focus attention on this specific cohort of patients, in order to describe in ever more detail any specific biomolecular aspects, and make full use of the pharmacological resources currently available.

DETAILED DESCRIPTION:
The definition "adolescent and young adults (AYA)" covers a broad group of patients ranging from the upper limit of the paediatric competence to the youngest patients usually considered and treated as adults. However, a well-defined and universally accepted age range is still not established. In fact, AYA includes patients from 16 to 24 years old according to the Britannic association "Teenage Cancer Trust" or 39 years old for the American National Cancer Institute definitions, respectively. Over the past 30 years, the incidence of cancer in AYA patients has increased globally by approximately 30%, estimating, in 2020 in U.S, 89,500 new cases and 9,270 deaths due to cancer among AYAs. Although the most frequent tumors are germ cell cancer for males and breast and thyroid cancers for female across the world, and confirmed also in Italian registries (https://www.aiom.it/wpcontent/uploads/2020/10/2020_Numeri_Cancro-operatori-web.pdf), malignancies arising from the gastrointestinal tract account all together for around 10% of cases. These are mainly represented by gastric cancer (up to 5%) followed by colorectal, neuroendocrine and hepatobiliary tumors.

Due to the high impact in terms of social impairment, a new and specific classification system based on the International Classification of Diseases for Oncology (ICD-O) and the World Health Organization (WHO) Classification of Tumors series for AYA cancers has been recently presented in order to sharpen the medical needs of this population.

However, AYA cohort remains a major clinical challenge, especially because of its poor representation in clinical trials, which prevent from the possibility to create a profile with specific molecular and etiopathogenetic features. Even though a significant part of these tumors rises from a hereditary basis (often in patients already followed by medical Genetic Unit), in most cases, cancers are sporadic, only partially associated to earlier exposure to carcinogenic factors such as alcohol and smoking, as well as a sedentary lifestyle and poor dietary education. Therefore, many questions remain unsolved regarding carcinogenesis, treatment, prognosis, and, eventually, prevention for family members of these patients.

Moreover, AYAs have a higher risk - even if lower than pediatric patients - to present long-term and late-onset side effects, concerning infertility, sexual disfunction, cardiotoxicity and second tumors. Early predictors biomarkers of these potential consequences are strongly needed. Considering current scarce information regarding how to improve outcomes of young patients affected by GI cancers and neuroendocrine neoplasms, this study aims to shed light on the biological behavior and the unmet needs of this population, by correlating clinical and biological factors to clinical outcomes. The main goal will be, firstly, the creation of a common and unique platform for acquiring biological samples and subsequently, potentially the identification of predictive and prognostic biomarkers.This study comprises both a retrospective and prospective phase. For the retrospective one, AYA patients will be included with GI or NeuroEndocrine (NE) malignancies (histologically confirmed). In the prospective part, when the study will be actively recruiting, clinical and biological data of all AYA patients will be collected and analyzed, according to specific outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age at diagnosis from18 to 39 years of age
* Carcinoma (without limitations for histologic subtypes) from any primary sites: esophagus, stomach, pancreas, biliary tract, liver, small bowel, colon, rectum, anus and cancer of unknown origin
* Neuroendocrine neoplasm (NEN) from Gastroenteropancreatic GEP or lung/thymus origin
* Tumors at any stage at the first visit
* Tumors of any grade
* Histological diagnosis obtained within two years from the time of enrollment or willingness to undergo bioptic procedure for diagnosis

Exclusion Criteria:

* Age at diagnosis > 39 years old

Ages: 18 Years to 39 Years | Sex: All
Age Groups: Adult
Study Population: young adults (18-39 years) with gastrointestinal and neuroendocrine tumors at any stage and any grade with histological diagnosis obtained within two years from the time of enrollment or willingness to undergo bioptic procedure for diagnosis
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Numbers of partecipants with genetic alterations | 3,5 years
  Prospective and retrospective observational study to analyze the frequency of tumors in young adults (18-49 years) with gastrointestinal and neuroendocrine tumors. Identification of genetic alterations with correlation between somatic and germline alterations.

SECONDARY OUTCOMES:
Number of partecipants with survival outcomes | 3,5 years
  Describe survival outcomes (overall survival and progression-free survival) according to the main clinical-pathological features and treatment received.
Number of partecipants toxicities | 3,5 years
  Describe potential toxicities developed as results of treatments according to clinical-pathological, genomic features and treatment received.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Spada, MD, Principal Investigator — Istituto Europeo di Oncologia
Locations (1):
- European Institute of Oncology, Milan, Italy

IPD SHARING:
Plan to Share IPD: No